CLINICAL TRIAL: NCT04179643
Title: Phase 1 Open Label, Dose Escalation Trial of Intracoronary Infusion of AB-1002 in Subjects With NYHA Class III Heart Failure
Brief Title: AB-1002 in Patients With Class III Heart Failure
Acronym: NAN-CS101
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AskBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NAN-CS101
Record Dates: First submitted 2019-09-06; First posted 2019-11-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Congestive Heart Failure; Heart Failure; Heart Disease, Ischemic; Cardiovascular Diseases; Heart Failure, Systolic; Heart Failure，Congestive; Heart Arrhythmia; Heart Failure, Diastolic; Heart; Complications
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia; Cardiovascular Diseases; Heart Failure, Systolic; Arrhythmias, Cardiac; Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 3.25E13vg AB-1002 (Experimental): Intracoronary Infusion of 3.25E13vg AB-1002 up to 6 subjects
  Interventions: Biological: 3 x 10e13vg AB-1002
- 1.08E14vg AB-1002 (Experimental): Intracoronary Infusion of 1.08E14vg AB-1002 to 6 subjects
  Interventions: Biological: 3 x 10e13vg AB-1002
- PLN-R14Del patients: 3.25E13vg AB-1002 (Experimental): Intracoronary Infusion of AB-1002 at 3.25E13vg up to 6 subjects with PLN-R14Del genetic mutation
  Interventions: Biological: 3 x 10e13vg AB-1002

INTERVENTIONS:
Biological: 3 x 10e13vg AB-1002 — There are 2 components to AB-1002. The first is an active I-1 transgene (AA 1-65 with T35D), and the second is the vector, BNP116, which delivers the gene selectively to the heart after intracoronary administration.

SUMMARY:
This is a Phase 1, prospective, multi-center, open-label, sequential dose escalation study to explore the safety, feasibility, and efficacy of a single intracoronary infusion of AB-1002 in patients with NYHA Class III heart failure. Patients with non-ischemic cardiomyopathy will be enrolled until up to 17 subjects have received infusions of investigational product. All patients will be followed until 12 months post treatment intervention, and then undergo long-term follow-up via semi-structured telephone questionnaires every 6 months for an additional 24 months (+/- 30 days).

DETAILED DESCRIPTION:
The safety endpoints will be assessed over the 12-month follow-up period

* Adverse Events
* Clinical laboratory tests
* Vital signs
* Electrocardiograms

Efficacy Endpoints

The efficacy endpoints assessed from baseline to 6 and 12 months will include the following:

* Observed and changes from baseline in peak VO2 assessed by cardiopulmonary exercise testing
* Observed and changes from baseline in 6-minute walk test
* Observed and changes from baseline in NYHA Classification
* Total number of days alive out-of-hospital

The secondary efficacy endpoints will explore efficacy. Functional endpoints will be assessed as changes from baseline to 6 and 12 months following investigational product administration as indicated. These endpoints include:

Functional Status & Hospitalizations

* Peak VO2 assessed by cardiopulmonary exercise testing
* 6-minute walk test
* New York Heart Association (NYHA) Classification
* Total number of days alive out-of-hospital (as well as total days out-of-hospital as a % of total days alive post study intervention)

Physiologic Assessments at 6 and 12 months compared to baseline

* Echocardiographic assessments of LVEF, LVEVD, LVEDVI, VLESV, LVEVI, SpI and GLSand degree of mitral regurgitation
* NT-proBNP level

Quality of Life at Week 8, 6 and 12 months compared to baseline

o Health related quality of life as assessed by Minnesota Living with Heart Failure Questionnaire (MLWHFQ) and Kansas City Cardiomyopathy Questionnaire

The following endpoints will also be measured over the 12 month follow-up period and long-term follow-up period (until month 36 post-intervention):

* Survival
* Cardiac transplantation
* Left ventricular assist device (LVAD) implantation

ELIGIBILITY:
Inclusion criteria:

* Age >18 years of age
* Chronic non-ischemic cardiomyopathy
* LVEF 15% ≤ 30% by transthoracic echocardiography (TTE) within 6 months prior to enrollment
* NYHA Class III HF for a minimum of 3 months HF despite appropriate medical therapy (defined below):

  * Treatment with appropriate HF therapy as tolerated, including, but not limited to:
  * Beta blocker therapy and angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) or sacubitril/valsartan combination therapy (Entresto) for ≥ 90 days prior to enrollment. May also receive aldosterone antagonist therapy. Doses of the above medications must be stable for ≥ 30 days prior to enrollment; and
  * Cardiac resynchronization therapy (CRT), if clinically indicated, must have been implanted ≥ 90 days prior to enrollment. Internal cardioverter defibrillator (ICD) must be implanted, if clinically indicated ≥ 30 days prior to enrollment
* Females of childbearing potential must use at least one of the following acceptable birth control methods throughout the study and for 6 months after IP administration:
* Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum prior to IP administration
* Intrauterine device in place for at least 90 days prior to receiving IP
* Barrier methods (diaphragm plus spermicide or condom) starting at least 30 days prior to receiving IP
* Abstinence (the subject must be willing to remain abstinent from screening to 6 months after receiving IP). Females are allowed to claim abstinence as their method of contraception only when it is the preferred and usual lifestyle of the subject
* Surgical sterilization of the partner(s) (vasectomy) for >180 days prior to IP administration
* Hormonal contraceptives starting > 90 days prior to IP. If hormonal contraceptives are started less than 90 days prior to receiving IP, subjects must agree to use a barrier method (diaphragm plus spermicide or condom) from screening through 90 days after initiation of hormonal contraceptives
* Males subjects capable of fathering a child:
* Must agree to use a condom from IP administration through 6 months after the time of IP administration
* Must agree not to donate sperm for 6 months after time of receiving IP
* Documented evidence of vasectomy in males for 180 days minimum prior to receiving IP is an acceptable form of contraception
* Males who claim abstinence as their method of contraception are allowed provided they agree to use barrier methods should they become sexually active from screening through 6 months after receiving IP. Males are allowed to claim abstinence as their method of contraception only when it is the preferred and usual lifestyle of the subject
* Ability to sign Informed Consent Form (ICF) and Release of Medical Information Form
* Appropriate candidate for protocol-specified intracoronary infusion in the judgment of the infusing interventional cardiologist

Cohort 3: medical history documentation of PLN-R14Del mutation and an ICD in situ (at least 30 days prior to enrollment)

Exclusion Criteria:

* Chronic ischemic cardiomyopathy
* Intravenous (IV) inotropic therapy, intra-aortic balloon pump (IABP) or percutaneous cardiac assist device therapy within 30 days prior to enrollment
* Restrictive cardiomyopathy, obstructive cardiomyopathy, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease, or dyskinetic LV aneurysm
* Cardiac surgery or percutaneous coronary intervention (PCI) within 30 days prior to enrollment
* Third degree heart block
* Clinically significant myocardial infarction (MI) in the judgment of the subject's physician (e.g., ST elevation MI [STEMI] or large non-STEMI) within 6 months prior to enrollment
* Prior heart transplantation, left ventricular reduction surgery (LVRS), cardiomyoplasty, passive restraint device (e.g., CorCap™ Cardiac Support Device), surgically implanted LVAD or cardiac shunt
* Likely to receive cardiac resynchronization therapy, cardiomyoplasty, LV reduction surgery, heart transplant, conventional revascularization procedure, or valvular repair within 3 months of IP dosing
* Known hypersensitivity to contrast dyes used for angiography; history of, or likely need for, high-dose steroid pretreatment prior to contrast angiography
* Expected survival < 1 year in the judgment of the investigator
* Active or suspected infection within 48 hours prior to enrollment as evidenced by fever or positive culture
* Known intrinsic liver disease (e.g., cirrhosis, hepatitis A, chronic hepatitis B or hepatitis C virus infection). If serology is positive and PCR is negative, subject may be eligible (confirm with medical monitor).
* Liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase) > 2x upper limit of normal (ULN) within 30 days prior to enrollment.
* Renal Failure, dialysis dependent or serum creatinine > 2.5 mg/dl within 30 days prior to enrollment
* Bleeding diathesis or thrombocytopenia defined as platelets <50,000 platelets/μL within 30 days prior to enrollment
* Anemia defined as hemoglobin <10 g/dL or transfusion dependent within 30 days prior to enrollment
* Neutropenia defined as absolute neutrophils <1500 mm3 within 30 days prior to enrollment
* Known AIDS or HIV-positive status, or a previous diagnosis of immunodeficiency with an absolute neutrophil count <1000 cells/mm3
* Previous participation in a study of gene transfer
* Receiving investigational intervention or participating in another clinical study within 30 days or within 5 half-lives of another investigational drug administration prior to administration of NAN-101 that may impact the therapeutic potential of NAN-101.
* Pregnancy or breastfeeding at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Observed and change from baseline in Peak VO2 | Measured at screening, month 6, 9 and month 12
  Cardiopulmonary exercise testing using a modified Bruce protocol
Observed and change from baseline in Echocardiographic assessment in Left Ventricular Ejection Fraction | Measured at screening, 18-24 hours post intervention, week 4, Month 3, Month 6 and Month 12
  Echocardiography LVEF measurement

SECONDARY OUTCOMES:
Observed and change from baseline in 6-minute walk test distance | Measured at screening, Month 3, Month 6 and month 12
  Analysis of Percent predicted in heart failure subjects compared to normal subjects

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Minneapolis Heart Foundation Institute, Minneapolis, Minnesota
  - The Linder Center for Education and Research at The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Wisconsin at Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henry TD, Chung ES, Alvisi M, Sethna F, Murray DR, Traverse JH, Roessig L, Roberts L, Reddy S, Chen Y, Ozkan TG, Webb S, Mittal M, Ervin L, Sadek H, Mikhail S, Haghighi K, Jiang C, Samulski RJ, Kranias EG, Tretiakova AP, Hajjar RJ. Cardiotropic AAV gene therapy for heart failure: a phase 1 trial. Nat Med. 2025 Nov;31(11):3845-3852. doi: 10.1038/s41591-025-04011-z. Epub 2025 Oct 21. PMID 41120766